CLINICAL TRIAL: NCT05837884
Title: Predicting Progression of Developing Myeloma in a High-Risk Screened Population and General Population
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PROMISE-ISRAEL
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-degree relative of a patient with a plasma cell dyscrasia or another blood cancer.: Individuals will ensure they are eligible by filling out an eligibility questionnaire confirming they meet all eligibility criteria. Individuals will provide informed consent to complete the baseline questionnaire and provide a blood sample that will be used to determine whether they have a monoclonal protein
  Interventions: Diagnostic Test: blood sampling
- Control group: The individuals without a relative of a patient with a plasma cell dyscrasia or another blood cancer.
  This group will undergo the same procedures as the first-degree participants and these data will be used for comparison between the populations.
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — Participants will provide a blood sample that will be used to determine whether they have a monoclonal protein

SUMMARY:
We will seek consent from participants to use the data and biospecimens collected according study protocol to address additional research questions for MGUS, SMM, MM, and other conditions.

Our overarching hypothesis is that early detection of MGUS/SMM in a high- risk population, along with the comprehensive characterization of genomic/epigenomic and microenvironmental/immune regulators of disease progression will lead to strategies that intercept disease progression and improve survival.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a plasma cell dyscrasia characterized by bone marrow (BM) infiltration and lytic bone lesions. Over 30, 000 Americans are diagnosed annually with MM. The estimated US prevalence is rising, and this trend is likely to continue due to improvements in diagnosis and therapy. Despite recent advances in therapy, MM remains a fatal disease with a median survival of 5-10 years and most patients still succumb to disease progression. Although many patients are diagnosed with earlier phases of disease, most patients do not receive treatment until their disease progresses, at which time they have overt end-organ damage. This concept of initiating therapy at the time of symptomatic disease is analogous to initiating therapy in patients with solid tumors only after the development of measurable metastatic disease. It is therefore not surprising that cure is not achieved for most patients with MM.

Recent studies have shown that MM is consistently preceded by MGUS and SMM. The incidence of MGUS is about 3% of the general population aged 50 years. This was through the analysis of a cohort of 77,000 people enrolled in a prospective population-based cancer screening trial that showed that multiple myeloma is consistently preceded by a precursor MGUS state. MGUS progresses to over MM at a slow rate of 1% per year, but in some patients, the risk may be as high as 58% in 20 years. SMM has an annual risk of progression of 10%. The rate of progression of high-risk SMM is as high as 70% in 5 years.

MGUS and SMM are often diagnosed incidentally when a physician orders a serum protein electrophoresis (SPEP) for a differential diagnosis of anemia, bone pain or renal insufficiency. Screening for early cancer detection has been implemented for many cancers including breast cancer (with mammography) and colon cancer (with colonoscopy) with variable success. However, a simple blood test for SPEP can accurately diagnose the presence of a plasma cell dyscrasia, indicating that early detection can identify these precursor conditions. In addition, recent studies have demonstrated that early detection of MGUS can lead to improved overall survival compared to incidental diagnosis of overt myeloma, presumably because these patients are followed more carefully and receive treatment before end-organ damage develops.

Therefore, high-risk populations include individuals with a first-degree relative that has been diagnosed with a plasma cell dyscrasia or other hematologic malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Must meet criteria of the high-risk population as described with one of the below criteria

  * ≥ 30 years AND
  * first-degree relative of a patient with a plasma cell dyscrasia such as MGUS, SMM, MM, and Waldenström's Macroglobulinemia, or another blood cancer.

OR

* Age ≥ 18 years with 2 or more first- or second-degree relatives with a plasma cell dyscrasia such as MGUS, SMM, MM, and Waldenström's Macroglobulinemia, or another blood cancer '
* Voluntary written informed consent must be given with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care

Exclusion Criteria:

* • Persons diagnosed with cancer at any site (including hematologic cancers) with symptomatic disease requiring active therapy.

  * Persons with an already diagnosed plasma cell dyscrasia such as MGUS, SMM, MM, and Waldenström's Macroglobulinemia
  * Female patient who have a positive serum pregnancy test during the screening period or a positive pregnancy test.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals who are first-degree relatives of hematological patients and A control group of healthy individuals who are not related to hematological patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence and Incidence | Every individual will have a different duration throughout the study depending on their diagnosis.
  Prevalence and Incidence of Monoclonal gammopathy of undetermined signiificance (MGUS)/smoldering multiple myeloma (SMM) in a high-risk population of family history positive individuals

SECONDARY OUTCOMES:
Presence of clinical alterations | Every individual will have a different duration throughout the study depending on their diagnosis.
  one of the objectives of the trial is to determine clinical alterations present in individuals with monoclonal gammopathies who are diagnosed through screening of a high- risk population.
Determination of natural history of screen-detected vs. incidentally detected MGUS/SMM | Every individual will have a different duration throughout the study depending on their diagnosis.
  One of the objectives of the trial to determine the natural history of screen-detected vs. incidentally detected MGUS/SMM. The present study of screened-detected MGUS/SMM can be compared to Dana-Farber Cancer Institute, Department of Hematologic Malignancies cohort of MGUS/SMM individuals incidentally diagnosed and longitudinally followed.
Determination clinical and epidemiological risk factors | Every individual will have a different duration throughout the study depending on their diagnosis.
  One of the objectives of the trial to determine the clinical and epidemiological risk factors for progression of MGUS/SMM to MM in a high-risk population of family positive cases.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Soroka, Beersheba
  - Rabin medical center, Petah Tikva
  - TASMC, Tel Aviv

IPD SHARING:
Plan to Share IPD: No